CLINICAL TRIAL: NCT05534477
Title: Verily Clinical Study Watch Analytical Validation Study
Status: Active, not recruiting | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 104126
Record Dates: First submitted 2022-08-23; First posted 2022-09-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy Population; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Verily Clinical Study Watch — The Study Watch is an investigational wrist worn wearable device made with biocompatible contact materials containing various sensors capable of continuous recording of physiological, activity, and environmental data.
Device: Vivalink ECG Patch — The Vivalink ECG Patch is a continuously recording ECG monitor and will be used as a reference device for measuring participants' pulse rate, pulse rate variability, and pulse rate coverage. The Vivalink ECG Patch is a medical device manufactured by VivaLNK Inc. and has been cleared by the FDA.
Device: Modus StepWatch 4 — Modus StepWatch 4 is an ankle-worn wearable medical device, and will be used as a reference device for measuring participants' ambulatory time and daily step count. The Modus StepWatch 4 is FDA listed.

SUMMARY:
This study is designed to evaluate the performance of the Verily Clinical Study Watch for the quantification of participants' movement and pulse rate when the wearer is at rest.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 22 and ≤ 80 years old
* Participant understands the study requirements and is able and willing to provide written informed consent
* Participant is without significant limitation in ability to participate in the study, in the opinion of the investigator
* Participant owns a smartphone with a data plan and be the primary user of the smartphone; smartphone must be compatible with the applications used in the study
* Participant is a US Resident

Exclusion Criteria:

* Participant has tremor or significant life-threatening arrhythmia
* Participant is allergic to nickel or metal jewelry
* Participant has a known severe allergy to polyester, nylon, or spandex
* Participant has a known allergic reaction to adhesives or hydrogels
* Participant has a tattoo covering the area where the watch face would rest on either wrist
* Participant has planned international travel during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 100 participants will be enrolled. This is a decentralized study across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of pulse rate when wearer is at rest | Approximately 14-day at-home observational period with two virtual visits, one at the beginning and the other at the end of the at-home period.
  To evaluate the accuracy of the Verily Clinical Study Watch's ability to measure pulse rate when wearer is at rest during unsupervised free-living conditions. Pulse rate measurements will be compared against heart rate output from the reference device (FDA cleared ECG patch).
Sensitivity of movement detection | Approximately 14-day at-home observational period with two virtual visits, one at the beginning and the other at the end of the at-home period.
  To evaluate the accuracy of the Verily Clinical Study Watch's ability to detect movement (rest vs not rest) during supervised conditions. Movement detection will be compared against virtual supervised observer-reference labels of rest vs not rest.
Specificity of movement detection | Approximately 14-day at-home observational period with two virtual visits, one at the beginning and the other at the end of the at-home period.
  To evaluate the accuracy of the Verily Clinical Study Watch's ability to detect movement (rest vs not rest) during supervised conditions. Movement detection will be compared against virtual supervised observer-reference labels of rest vs not rest.

CONTACTS AND LOCATIONS:
Overall Officials: Scooter Plowman, MD, Principal Investigator — Verily Life Sciences
Locations (1):
- Verily Life Sciences, South San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No